CLINICAL TRIAL: NCT06131853
Title: Physical Activity, Fear of Falling, Fatigue and Functionality in Prostate Cancer
Brief Title: Kinesiophobia in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Asst Prof Dr, Selcuk University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023/11.09
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer; Kinesiophobia; Physical Inactivity
MeSH Terms: conditions — Prostatic Neoplasms; Kinesiophobia; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prostate group (Experimental)
  Interventions: Other: survey evaluation
- control group (Active Comparator)
  Interventions: Other: survey evaluation

INTERVENTIONS:
Other: survey evaluation — assessment of physical activity, fatigue, fear of movement, and quality of life

SUMMARY:
This study aimed to investigate the effects of prostate cancer on patients' physical activity, kinesiophobia, fatigue and functionality.

This research is a prospective study to be conducted on volunteer individuals between the ages of 40-75. People diagnosed with prostate cancer (study group) and healthy adults who have not been diagnosed with prostate cancer before (control group) will be included in the study. The demographic characteristics, physical activity levels and quality of life of all individuals participating in the study will be evaluated with an online form. In demographic data, physical, sociodemographic data such as age (years), height (cm), body weight (kg), body mass index (kg/m2) and disease-specific information will be recorded. Physical activity level will be measured with the International Physical Activity Survey short form (UFAA), fatigue with the Functional Evaluation of Chronic Disease Treatment-Fatigue Questionnaire, fear of movement with the Causes of Fear of Movement Questionnaire, and quality of life with the Functional Evaluation of Cancer Treatment-Prostate Version questionnaire (KHTFD-Y).

ELIGIBILITY:
Inclusion Criteria:

* (for prostate cancer-study group)

  * Being between the ages of 40-75
  * Want to participate in the study
  * Being able to read and write
  * Being diagnosed with prostate cancer by a specialist physician,
  * Being able to provide their mobility independently,
* (for healthy controls - control group)

  * Being between the ages of 40-75
  * Not having any previous cancer history and not having undergone cancer surgery
  * Volunteering to participate in the study

Exclusion Criteria:

* Those with a previously known or accompanying diagnosis of dementia
* Not wanting to participate in the study
* The individual has a disease that may prevent him or her from understanding and completing the survey.
* Illiterates
* Those who do not want to participate in the research voluntarily
* Having active metastasis
* Having undergone chemotherapy and radiotherapy in the last 6 months

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Survey short form | 10 minutes
  The short form consists of 7 questions. The form provides information about the frequency and time spent in walking, moderate physical activity, and vigorous physical activity.
Functional Assessment of Fatigue Chronic Disease Treatment-Fatigue Questionnaire | 10 minutes
  It consists of 13 questions that evaluate the level of fatigue that occurred during daily activities in the last 7 days. Scoring varies between 0-52. High scores indicate less fatigue.
Reasons for Fear of Movement Questionnaire | 10 minutes
  It allows the causes of kinesiophobia to be identified and both biological and psychological causes to be determined separately. The average of the scores obtained from the biological and physiological subscales gives the total score from the survey. A 5-point Likert scoring (1 = Totally disagree, 5 = Completely agree) is used in the scale. An individual's high score from the survey indicates that he/she has more fear of movement.
Functional Evaluation of Cancer Treatment-Prostate Version questionnaire | 10 minutes
  It consists of 13 questions that evaluate the level of fatigue that occurred during daily activities in the last 7 days. Scoring varies between 0-52. High scores indicate less fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)